CLINICAL TRIAL: NCT00588432
Title: Characterization of Skeletal Muscle Using Magnetic Resonance Elastography (MRE)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Kai-Nan An, May Clinic
Other Study IDs: 2391-02; 5R01EB000812 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Stroke; Immobilization; Myofacial Pain; Hyperthyroid Myopathy
Keywords: Stroke; Immobilization; Myofacial Pain; Hyperthyroid Myopathy
MeSH Terms: conditions — Stroke; Facial Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- 1: Hemiparesis as the result of an ischemic hemispheric stroke.
- 2: Immobilization following severe Achilles tendon tear or rupture, ankle injury or plantar fascial pain.
- 3: Myofascial trigger points in trapezius muscle.
- 4: Hyperthyroid Myopathy

SUMMARY:
The goal of this proposal is two-fold: (1) to further develop and validate a technology, magnetic resonance elastography (MRE), for quantitatively imaging mechanical properties and tension distribution in muscle and (2) to apply the technique for in vivo evaluation of patients with four common, and clinically significant muscle disorders (spasticity, disuse atrophy, myofascial pain and a metabolic myopathy). These studies will employ a magnetic resonance imaging sequence with synchronous motion-sensitizing gradients to map propagating shear waves in the muscle. The technique will assess the mechanical properties of the muscle and its tension distribution. Specifically, the study can be divided into three specific aims. Aim 1: Optimize MRE methods of acquisition and analysis for the assessment of muscle, including electromechanical drivers, data acquisition techniques, and methods for image analysis. Advanced techniques for very rapid MRE assessment of muscle will continue to be developed. Aim 2: Validate the MRE assessment of muscle properties and tension with phantom, ex-vivo muscle, and Finite Element Modeling (FEM) techniques. Finite Element Analysis will be performed by using both phantom and bovine muscles to better correlate MRE wave-length findings as function of muscle properties, tension and fiber architecture. Aim 3: Study In Vivo Normal and Abnormal Muscle. The MRE technique will be applied in vivo to provide elastographic images of abnormal muscle with known disorders. The patient groups chosen for study are each important in their own right, and furnish unique information across the spectrum of muscular disease and dysfunction. Groups to be studied include individuals with new onset of spasticity following an ischemic, hemispheric stroke, disuse atrophy as a result of immobilization, metabolic (hyperthyroid) myopathy and myofascial pain for trigger point identification. The overall hypothesis of this work is that will bring benefits to both basic research and clinical care.

ELIGIBILITY:
Inclusion Criteria:

Normals:

* Healthy individuals

Stroke:

* a first stroke (i.e., a unilateral, ischemic hemispheric stroke) within the previous one to two months, ability to cooperate and follow simple commands, and gastrocsoleous strength in the affected lower extremity of between trace and 50% of normal.

Immobilization:

* immobilized in a cast (typically 6 weeks) following sugical repair of a severe Achilles tendon tear or rupture, ankle injury or plantar fascial pain

Myofascial Pain:

* history of pain in trapezius confirmed by clincal examination. The examiner will perform snapping palpation over the MFTP. If a localized, transient contraction is observed, the response is considered to be positive and the subject will be considered eligible for entry into the study.

Hyperthyroid Myopathy:

* clinical assessment in combination with a serum hormone profile of increased Free Thyroxine (FT4) and Triiodothyronine (T3) in the face of suppressed levels of Thyroid Stimulating Hormone (TSH).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of the community and patients of the study investigators.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2003-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States